CLINICAL TRIAL: NCT06303297
Title: Combined Effects of Reflexology and Generalized Stretching on Insomnia, Vasomotor Symptoms and Quality of Life in Postmenopausal Females
Brief Title: Effects of Reflexology and Generalized Stretching in Postmenopausal Females.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0576
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Postmenopausal Disorder
Keywords: Female; insomnia; postmenopausal; quality of life; reflexology
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REFLEXOLOGY (Experimental)
  Interventions: Other: REFLEXOLOGY
- GENERALIZED STRETCHING (Active Comparator)
  Interventions: Other: GENERALIZED STRETCHING

INTERVENTIONS:
Other: REFLEXOLOGY — will receive foot and hand reflexology and stretching. The researcher will administer foot and hand reflexology to the participant for a period of 3 weeks this last for a duration of 10 min on each hand and foot with total duration of 40 minutes. Foot reflexology include general foot massage, including the foot rotation, Achilles stretching, and the foot extension and stretching, will be performed for a minute on each foot. In the right foot, the bottom of the heel will be kept with the left hand, and the metatarsal arch of the same foot will be held with the other hand. Then, the foot will be rotated clockwise and counter clockwise three times each direction. The same technique will be performed on the left foot. On hand lubricated with moisturizer to the dorsal and plantar surface and apply pressure on for 10 minutes. Noninvasive and safe complementary therapy that involves a direct pressure on specific body points connecting specific organs.
  Arms: REFLEXOLOGY
Other: GENERALIZED STRETCHING — will receive Stretching of upper and lower limbs. The stretching program lasts for 3 weeks with 60 min of stretching session 3 times a week. Extension of body include shoulder extension, torso rotation, hip extension, calf stretching (ankle pumps). ten stretches of 30 s each, with 15 s of rest between each stretch
  Arms: GENERALIZED STRETCHING

SUMMARY:
To determine the combined Effects of reflexology and generalized stretching on insomnia, vasomotor symptoms and quality of life in postmenopausal females

ELIGIBILITY:
Inclusion Criteria:

* BMI less than 30 kg/m2
* Residents of rural areas
* Stable vital signs
* Participants with natural cessation of menstrual periods for at least 12 months
* Moderate and severe hot flash

Exclusion Criteria:

* Participants with history of hysterectomy surgical menopause females
* Participants with orthopedic disorder
* Participants taking sleeping pills
* Women suffer from pathological conditions for example cardiac disease, cancer impaired skin integrity
* Participants with history of recent bone fracture
* Severe pathology(eczema) of feet

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — post partum females
Enrollment: 32 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Insomnia severity index score | 3rd week
  This questionnaire is a 7 items questionnaire which is used to assess sleep problems. It scoring is done through Likert type scale ranging from 0 to 4, where higher score represents higher sleep problem. Its score is range from 0 to 28 where 0 to 7 shows no clinically significant insomnia, 8 to 14 shows subthreshold insomnia, 15 to 21 shows moderate severity of insomnia and 22 to 28 shows severe severity of insomnia. It is a reliable and valid tool with internal consistency of 0.74 and correlation ranging from 0.36 to 0.54.
Menopause Rating Scale | 3rd week
  Menopause Rating Scale is a 11 items questionnaire which is use to assess vasomotor symptoms like hot flush, palpitations, sleep problem, bladder symptoms and other symptoms.
  Its score range is from 0 to 4, where 0 shows no complain and 4 shows severe symptoms. Its total score range is from 9 to 21, where higher the score higher are the symptoms. It has good validity and reliability. It has Cronbach alpha value of 0.86 and internal consistency of 0.81.
Menopause Specific Quality of Life | 3rd week
  Menopause specific quality of life (MENQOL) questionnaire is a 29 items questionnaire which is used to assess quality of life among menopausal women. It has further four domains vasomotor (item 1 to 3), sexual (item 27-29), psychosocial (item 4-10) and physical (item 11 to 26). It is a reliable and valid tool with Cronbach value of 0.70 and internal consistency of 0.45.

CONTACTS AND LOCATIONS:
Overall Officials: hina gul, Principal Investigator — Riphah International University
Locations (1):
- Akhtar Saeed trust hospital,, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vogazianou A. Anatomy and physiology of the female reproductive system. Advanced Practice in Endocrinology Nursing. 2019:739-52.
- [Background] Hoare BS, Mikes BA, Khan YS. Anatomy, Abdomen and Pelvis: Female Internal Genitals. 2025 Feb 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554601/ PMID 32119488
- [Background] Sochocka M, Karska J, Pszczolowska M, Ochnik M, Fulek M, Fulek K, Kurpas D, Chojdak-Lukasiewicz J, Rosner-Tenerowicz A, Leszek J. Cognitive Decline in Early and Premature Menopause. Int J Mol Sci. 2023 Mar 31;24(7):6566. doi: 10.3390/ijms24076566. PMID 37047549
- [Background] Talaulikar V. Menopause transition: Physiology and symptoms. Best Pract Res Clin Obstet Gynaecol. 2022 May;81:3-7. doi: 10.1016/j.bpobgyn.2022.03.003. Epub 2022 Mar 16. PMID 35382992
- [Background] Yeo JH, Kim MT. Association of weight, smoking, and alcohol consumption with age at natural menopause. J Women Aging. 2023 Jul-Aug;35(4):343-353. doi: 10.1080/08952841.2022.2050157. Epub 2022 Mar 21. PMID 35312401
- [Background] Kalhan M, Singhania K, Choudhary P, Verma S, Kaushal P, Singh T. Prevalence of Menopausal Symptoms and its Effect on Quality of Life among Rural Middle Aged Women (40-60 Years) of Haryana, India. Int J Appl Basic Med Res. 2020 Jul-Sep;10(3):183-188. doi: 10.4103/ijabmr.IJABMR_428_19. Epub 2020 Jul 11. PMID 33088741
- [Background] Ragasudha A, Minnu S, Kumar RS. Menopause Induced Depression, Anxiety, Quality of Life, Lack of Sleep in Women: An Overview. Journal of Drug Delivery and Therapeutics. 2021;11(6):319-23.